CLINICAL TRIAL: NCT00637195
Title: Evaluation of the Immunogenicity and Safety of a Commercially Available Vaccine When Co-administered With GlaxoSmithKline Biologicals' HPV Vaccine (580299) in Healthy Female Subjects.
Brief Title: Immunogenicity and Safety of a Commercially Available Vaccine Co-administered With GSK HPV Vaccine (580299)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111567; 2007-007876-41 (EudraCT Number)
Record Dates: First submitted 2008-02-28; First posted 2008-03-17 (Estimated); Results first posted 2009-12-18 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Infections, Papillomavirus; Papillomavirus Vaccines
Keywords: Human papillomavirus (HPV) vaccine; Hepatitis B; Cervical cancer; HPV; Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections; Hepatitis B; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18; Engerix-B

ARMS (2):
- Cervarix™ & Engerix™ Group (Experimental): Subjects received 3 doses of GSK Biologicals' HPV vaccine (580299) (Cervarix™) (Months 0, 1 & 6) and 4 doses of Hepatitis B (Engerix™) vaccine (Months 0, 1, 2 & 12).
  Interventions: Biological: Subjects received 3 doses of GSK Biologicals' HPV vaccine (580299) (Cervarix™); Biological: Engerix™
- Engerix™ Group (Active Comparator): Subjects received 4 doses of Hepatitis B (HBV) vaccine (Months 0, 1, 2 & 12).
  Interventions: Biological: Engerix™

INTERVENTIONS:
Biological: Subjects received 3 doses of GSK Biologicals' HPV vaccine (580299) (Cervarix™) — Intramuscular administration, 3 doses.
  Other Names: GSK Biologicals' HPV vaccine 580299
  Arms: Cervarix™ & Engerix™ Group
Biological: Engerix™ — Intramuscular administration, 4 doses.
  Other Names: GSK Biologicals' vaccine 103860

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the necessary cause of cervical cancer. The current Phase 3b study is designed to assess the immunogenicity and safety of a commercially available vaccine co-administered with GlaxoSmithKline Biologicals' HPV vaccine GSK580299 in healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A female between, and including, 20 and 25 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and history directed clinical examination before entering into the study.
* Subjects must not be pregnant.
* Subjects must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after each dose of vaccine. Administration of routine vaccines such as meningococcal, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccines up to 8 days before the first dose of study vaccine is allowed.
* Concurrently participating in another clinical study, at any time during the study period (up to Month 13), in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* A subject planning to become pregnant, likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive precautions during the study period and up to two months after the last vaccine dose.
* Pregnant or breastfeeding women.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period
* Previous administration of components of the investigational vaccine.
* Previous vaccination against hepatitis B or planned administration of any hepatitis B vaccine other than that foreseen by the study protocol during the study period.
* History of hepatitis B infection.
* Known exposure to hepatitis B within the previous 6 weeks.
* Known acute or chronic, clinically significant neurologic, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* Cancer or autoimmune disease under treatment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2008-03-11 (Actual); Primary Completion 2008-06-20 (Actual); Study Completion 2009-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, La Louvière

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=211

REFERENCES:
- [Background] Leroux-Roels G, Haelterman E, Maes C, Levy J, De Boever F, Licini L, David MP, Dobbelaere K, Descamps D. Randomized trial of the immunogenicity and safety of the Hepatitis B vaccine given in an accelerated schedule coadministered with the human papillomavirus type 16/18 AS04-adjuvanted cervical cancer vaccine. Clin Vaccine Immunol. 2011 Sep;18(9):1510-8. doi: 10.1128/CVI.00539-10. Epub 2011 Jul 6. PMID 21734063
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 111567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Started | 76 | 76
Completed | 73 | 75
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (1.51) | 22.1 (1.32) | 22.3 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 76 | 152
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroprotected Against Hepatitis B Following 3 Doses of Engerix
Description: A subject seroprotected against hepatitis B is a subject with anti-hepatitis B surface antigen (HBs) antibody titers greater than or equal to 10 milli-international units per milliliter (mIU/mL).
Time Frame: Month 3
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, in subjects with available data and who were negative for anti-hepatitis B core antigen (anti-HBc) before vaccination .
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 72 | 75
Participants | 70 | 73

2. Primary Outcome: Anti-hepatitis B Surface Antigen (HBs) Antibody Titers Following 3 Doses of Engerix
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as milli-international units per milliliter (mIU/mL).
Time Frame: Month 3
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, in subjects with available data and who were negative for anti-hepatitis B core antigen (anti-HBc) before vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 72 | 75
mIU/mL | 156.1 [83.7 to 291.3] | 146.2 [86.6 to 246.9]

3. Secondary Outcome: Number of Subjects Seroconverted for Anti-human Papilloma Virus 16 and 18 (Anti-HPV-16 and Anti-HPV-18) Antibodies
Description: Seroconversion is defined as the appearance of antibodies with titers greater than or equal to the predefined cut-off value in the serum of subject seronegative before vaccination.
  Cut-off values assessed include 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: Months 2 and 7
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, only for subjects receiving Cervarix™ vaccine and with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 68 | 0
Participants
  Anti-HPV-16, Month 2: number analyzed (Participants) | 62 | 0
  Anti-HPV-16, Month 2 | 62 |
  Anti-HPV-16, Month 7: number analyzed (Participants) | 61 | 0
  Anti-HPV-16, Month 7 | 61 |
  Anti-HPV-18, Month 2 | 68 |
  Anti-HPV-18, Month 7: number analyzed (Participants) | 67 | 0
  Anti-HPV-18, Month 7 | 67 |

4. Secondary Outcome: Anti-HPV-16/18 Antibody Titers
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
Time Frame: Months 2 and 7
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, only for subjects receiving Cervarix™ vaccine with available data.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 68 | 0
EL.U/mL
  Anti-HPV-16, Month 2: number analyzed (Participants) | 62 | 0
  Anti-HPV-16, Month 2 | 3497.2 [2902.3 to 4214.1] |
  Anti-HPV-16, Month 7: number analyzed (Participants) | 61 | 0
  Anti-HPV-16, Month 7 | 8725.2 [7105.7 to 10714.0] |
  Anti-HPV-18, Month 2 | 2775.6 [2306.5 to 3340.1] |
  Anti-HPV-18, Month 7: number analyzed (Participants) | 67 | 0
  Anti-HPV-18, Month 7 | 4664.4 [3709.9 to 5864.3] |

5. Secondary Outcome: Number of Subjects Seroconverted for Anti-hepatitis B (HBs) Antibodies
Description: Anti-HBs seroconversion is defined as the appearance [i.e. titer greater than or equal to the cut-off value of 3.3 milli-international units/milliliter (mIU/mL)] of anti-HBs antibodies in the sera of subjects seronegative (with titers below the cut-off value) before vaccination.
Time Frame: Months 2, 3 and 13
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, in subjects with available data and who were negative for anti-hepatitis B core antigen (anti-HBc) before vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 55 | 64
Participants
  Month 2 | 46 | 54
  Month 3 | 55 | 63
  Month 13: number analyzed (Participants) | 52 | 63
  Month 13 | 52 | 63

6. Secondary Outcome: Number of Subjects Seroprotected Against Anti-Hepatitis B (HBs) Antibodies Following 2 Doses of Engerix and After Completing the 4-dose Engerix Vaccination Course
Description: A subject seroprotected against Hepatitis B is a subject with anti-HBs antibody titers greater than or equal to 10 mIU/mL.
Time Frame: Months 2 and 13
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 72 | 75
Participants
  Month 2 | 63 | 65
  Month 13: number analyzed (Participants) | 69 | 74
  Month 13 | 69 | 74

7. Secondary Outcome: Anti-HBs Antibody Titers Following 2 Doses of Engerix and After Completing the 4-dose Engerix Vaccination Course
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as mIU/mL.
Time Frame: At Months 2 and 13
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 72 | 75
mIU/mL
  Month 2 | 34.4 [17.1 to 69.5] | 35.7 [18.9 to 67.1]
  Month 13: number analyzed (Participants) | 69 | 74
  Month 13 | 19888.4 [13042.6 to 30327.5] | 16927.5 [11854.1 to 24172.3]

8. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include injection site pain, redness and swelling.
  Data are presented across doses.
Time Frame: During the 7-day period following any vaccination
Population: Analysis was performed on the Total Vaccinated cohort, which consisted of all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 76 | 76
Participants
  Pain | 76 | 62
  Redness | 26 | 12
  Swelling | 26 | 10

9. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include injection site pain, redness and swelling.
  Data are presented across doses.
Time Frame: During the 7-day period following the 4th dose of HBV vaccine
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 74 | 75
Participants
  Pain | 36 | 44
  Redness | 8 | 13
  Swelling | 12 | 10

10. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, rash, temperature [axillary route, ≥ 37.5 degree Celsius (°C)] and urticaria.
  Data are presented across doses.
Time Frame: During the 7-day period following any vaccination
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 76 | 76
Participants
  Arthralgia | 9 | 10
  Fatigue | 49 | 52
  Gastro-intestinal symptoms | 24 | 31
  Headache | 49 | 42
  Myalgia | 28 | 33
  Rash | 3 | 5
  Temperature ≥ 37.5°C | 9 | 5
  Urticaria | 1 | 3

11. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: as for outcome 10
Time Frame: During the 7-day period following the 4th dose of HBV vaccine
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 74 | 75
Participants
  Arthralgia | 1 | 4
  Fatigue | 26 | 34
  Gastro-intestinal symptoms | 3 | 13
  Headache | 21 | 25
  Myalgia | 4 | 18
  Rash | 1 | 0
  Temperature ≥ 37.5°C | 3 | 0
  Urticaria | 0 | 0

12. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: Unsolicited adverse event covers any adverse event reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 30-day period following any vaccination
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 76 | 76
Participants | 56 | 47

13. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: as for outcome 12
Time Frame: During the 30-day period following the 4th dose of HBV vaccine
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 74 | 75
Participants | 20 | 22

14. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Up to study end (Month 13)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 76 | 76
Participants | 2 | 2

15. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions
Description: Medically significant conditions include adverse events (AEs) prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: Up to study end (Month 13)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Number analyzed (Participants) | 74 | 75
Participants | 37 | 32

ADVERSE EVENTS:
Time Frame: From Month 0 up to Month 13.
Arm/Group | Cervarix™ & Engerix™ Group | Engerix™ Group
Serious Adverse Events (participants affected / at risk) | 2/76 | 2/76
Other Adverse Events (participants affected / at risk) | 76/76 | 73/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix™ & Engerix™ Group (N=76) | Engerix™ Group (N=76)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Graves-Basedow's disease (Endocrine disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix™ & Engerix™ Group (N=76) | Engerix™ Group (N=76)
Pain at injection site (General disorders) | 76 | 62
Redness at injection site (General disorders) | 26 | 12
Swelling at injection site (General disorders) | 26 | 10
Arthralgia (General disorders) | 9 | 10
Fatigue (General disorders) | 49 | 52
Gastrointestinal symptom (General disorders) | 24 | 31
Headache (Gastrointestinal disorders) | 49 | 42
Myalgia (General disorders) | 28 | 33
Rash (General disorders) | 3 | 5
Temperature (General disorders) | 9 | 5
Headache (Nervous system disorders) | 12 | 13
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Dysmenorrhoea (Reproductive system and breast disorders) | 7 | 6
Cystitis (Infections and infestations) | 5 | 4
Nasopharyngitis (Infections and infestations) | 6 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Influenza like illness (General disorders) | 1 | 4
Pharyngitis (Immune system disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.